CLINICAL TRIAL: NCT01954992
Title: A Randomized Phase 3 Study of the Efficacy and Safety of Glufosfamide Compared With Fluorouracil (5-FU) in Patients With Metastatic Pancreatic Adenocarcinoma Previously Treated With Gemcitabine
Brief Title: Glufosfamide Versus 5-FU in Second Line Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eleison Pharmaceuticals LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP-GF-301
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: glufosfamide; 5-FU; metastatic pancreatic adenocarcinoma
MeSH Terms: interventions — beta-D-glucosylisophosphoramide mustard; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glufosfamide (Experimental): Glufosfamide: 4500 mg/m2 IV over 6 hours on Day 1 of each 21-day cycle
  Interventions: Drug: Glufosfamide
- 5-FU (Active Comparator): Fluorouracil (5-FU): 600 mg/m2 IV over 30 minutes on Day 1 of each week
  Interventions: Drug: Fluorouracil

INTERVENTIONS:
Drug: Glufosfamide — Glufosfamide: 4500 mg/m2 IV over 6 hours (¼ dose over 30 minutes, ¾ dose over remaining 5.5 hours) on Day 1 of each 21-day cycle.
  Arms: glufosfamide
Drug: Fluorouracil — Fluorouracil (5-FU): 600 mg/m2 IV over 30 minutes on Day 1 of each week
  Other Names: 5-FU
  Arms: 5-FU

SUMMARY:
The study is designed to assess whether glufosfamide provides additional survival benefit as compared to bolus 5-FU in patients with metastatic pancreatic cancer who have already progressed or failed therapy on a gemcitabine based first line regimen.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Pancreatic adenocarcinoma proven either by histology (surgical biopsy) or cytology (CT- or endoscopic-guided)
* Metastatic pancreatic cancer
* Disease progression during or after treatment with gemcitabine (alone or in combination with other agents; at regular, not radiosensitizing, doses)
* Measurable or nonmeasurable disease by RECIST criteria (at least one target or nontarget lesion)
* Recovered from reversible toxicities of prior therapy
* ECOG performance status 0-1
* All women of childbearing potential and all men must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) from entry into the study through 6 months after the last dose of chemotherapy
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee

Exclusion Criteria:

* More than one prior systemic therapy regimen for metastatic pancreatic cancer (radiosensitizing doses of 5-FU or gemcitabine at the time of initial radiotherapy do not count as a prior systemic therapy regimen)
* Hormonal therapy, radiation therapy, biologic therapy, chemotherapy or other systemic antitumor therapy for pancreatic cancer within 14 days prior to Cycle 1 Day 1
* Insulin-dependent diabetes mellitus (patients with type 2 diabetes controlled with oral glucose lowering agents and the occasional use of insulin are permitted in the study)
* Symptomatic brain metastases (baseline CT scan is not required in asymptomatic patients)
* Active clinically significant infection requiring antibiotics
* Known HIV positive or active hepatitis B or C
* Recent (one year) history or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4), particularly coronary artery disease, arrhythmias or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, or congestive heart failure
* No other active malignancies (other than treated non-melanoma skin cancer or treated in situ cancer) within the past year
* Major surgery within 3 weeks of the start of study treatment, without complete recovery
* Clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including electrolytes, and urinalysis)

  * Hemoglobin <9 g/dL (may receive transfusion or erythropoietin to maintain)
  * ANC <1500/μL
  * Platelet count <100,000/μL
  * Total bilirubin > 1.5×ULN
  * AST/ALT > 2.5-fold above ULN (>5-fold above ULN if liver metastases)
  * Phosphorus < LLN
  * Potassium < LLN
  * Serum creatinine > 2 mg/dL
  * Creatinine clearance < 60 mL/min (calculated by Cockcroft-Gault formula)
* Females who are pregnant or breast-feeding
* Participation in an investigational drug or device study within 14 days of the first day of dosing on this study
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study
* Any medical history, concurrent disease or concomitant medication which could reasonably predispose the patient to renal insufficiency while on study treatment
* Contraindication or unwillingness to undergo multiple CT scans
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2014-04; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Approximately 3-6 months
  Time from Randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Thomas, Study Director — Eleison Pharmaceuticals
Locations (3):
- United States (3):
  - Innovative Clinical Research Institute, Whittier, California
  - Moffitt Cancer Center, Tampa, Florida
  - Gabrail Cancer Center Research, Canton, Ohio